CLINICAL TRIAL: NCT04096391
Title: Post-market, Randomized, Controlled, Prospective Study Evaluating Intrathecal Pain Medication (IT) Versus Conventional Medical Management (CMM) in the Non-cancer, Refractory, Chronic Pain Population (PROSPER)
Brief Title: Post-market, Randomized, Controlled, Prospective Study Evaluating Intrathecal Pain Medication (IT) Versus Conventional Medical Management (CMM) in the Non-cancer, Refractory, Chronic Pain Population
Acronym: Prosper-001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evolve Restorative Center (Other)
Collaborators: Flowonix Medical (Industry); Celéri Health, Inc. (Industry); Advanced Infusion Solutions (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Prosper-001
Record Dates: First submitted 2019-09-12; First posted 2019-09-19 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Chronic Nonmalignant Pain; Pain, Intractable; Pain, Chronic
Keywords: Truncal Pain; Lower Extremity Limb Pain; Refractory Pain
MeSH Terms: conditions — Pain, Intractable; Chronic Pain | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1 ratio to one of two groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intrathecal Drug Delivery System (Active Comparator): Subjects randomized to the Intrathecal Drug Delivery System group will be implanted with the Prometra System under sterile technique in accordance with the Instructions for Use. The pump will be filled at the time of implantation with the prescribed medication.
  Interventions: Device: Flowonix Prometra® II Programmable Infusion System
- Conventional Medical Management (Active Comparator): Subjects randomized to the Conventional Medical Management group will continue with the standard of care procedures.
  Interventions: Drug: Pain Medicine

INTERVENTIONS:
Device: Flowonix Prometra® II Programmable Infusion System — The Flowonix Prometra® II Programmable Infusion System consists of an implanted infusion pump and catheter, and external components including a clinician programmer, refill and catheter access port kits, the PTC™(a subject operated controller).
  Arms: Intrathecal Drug Delivery System
Drug: Pain Medicine — Injections, spinal cord stimulation, peripheral nerve stimulation, pain medication, etc.
  Other Names: Systemic opioid therapy
  Arms: Conventional Medical Management

SUMMARY:
This study is being conducted to compare intrathecal morphine using the commercially available intrathecal drug delivery systems (IDDS), and conventional medical management (CMM) in subjects with non-cancer, refractory chronic pain.

DETAILED DESCRIPTION:
This study will evaluate the following objectives:

Primary objective:

1. To compare the change in pain intensity from baseline based on the Numeric Rating Scale [NRS] between subjects randomized to the IDDS group and subjects randomized to the CMM group.The comparison will be conducted at 3, 6, 9 and 12 months following enrollment. The evaluation at 6 months will be considered the primary time point for evaluation.

Secondary objectives:

For each of the following secondary objectives, the comparisons between the IDDS group and CMM group will be made using the intra-subject change from baseline as the dependent variable.

1. Compare the subject reported PROMIS 29 between the IDDS group and CMM group. Individual subject scores recorded at baseline and months 3, 6, 9 and 12.
2. Compare the accrued cost of therapy for pain control including those related to adverse events, ED visits, cost of medications between the IDDS group and CMM group
3. Compare the number of other concurrent treatments performed on each subject between the IDDS group and CMM group. Individual subject counts recorded at months 3, 6, 9 and 12 will be compared.

Additional safety objective:

1. To characterize pain and device related adverse events for all subjects throughout the study through completion of 12 month follow-up or subject exit.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have signed and dated the IRB approved Informed Consent Form and HIPAA Authorization prior to any study procedures being performed
2. Subject must be willing and able to complete study requirements including diaries, questionnaires and attend all visits, in the opinion of the investigator
3. Subject must be male or female and at least 22 years of age
4. Subjects who are female are non-lactating and if of childbearing potential have a negative urine pregnancy test at screening
5. Subjects who are currently be receiving ≤ 90 mg/day morphine per day dose (or MME), with stable dose at equivalent of systemic opioids at Screening
6. Subjects who are on a stable dose of opioids (no change in type or prescribed frequency or dose) for 30 days prior to the screening as documented in medical history;
7. Subjects who have refractory pain despite failure of regional minimally invasive treatment options, including epidurals, facets, rhizotomies, direct or indirect spinal stenosis treatments, etc.
8. Subjects who are a new candidate for chronic intrathecal drug therapy (including no prior intrathecal/epidural trial for pump infusion therapy)
9. Subjects have not been implanted with a spinal cord stimulator for pain
10. Subjects currently do not have an implanted spinal cord stimulator for pain
11. Subjects who have a diagnosis of nonmalignant, chronic intractable pain as documented in the medical history
12. Subjects who are medically stable and able to undergo surgery for implantation of the Prometra® II Infusion System
13. Subject must have completed a psychological evaluation within 6 months prior to Screening
14. Subject must complete an intrathecal trial resulting in candidacy for pump implantation during Screening

Exclusion Criteria:

A potential subject who has any contraindications listed in the Prometra® II labeling or any contraindications of intrathecal agents employed in the United States within the PACC, will be excluded. All subjects meeting any of the following criteria will also be excluded from this study:

1. Subjects currently have a spinal cord stimulator implanted for pain
2. Subjects previously had a spinal cord stimulator implanted for pain
3. Subjects who have psychological or other health conditions, financial, and/or legal concerns (within 3 months prior to Screening) that would interfere with the subject's ability to fulfill the requirements of the protocol as per the investigator's opinion
4. Subjects who have a history of alcohol abuse or illicit drug use within 2 years of screening
5. Subjects who have an active malignancy or has been diagnosed with cancer and has not been in remission for at least 1 year prior to Screening
6. Subjects who are female and who are pregnant, nursing or planning a pregnancy during the study or females of childbearing potential who are unable or unwilling to use a form of contraception during the study.
7. Subjects who plan to enroll or is currently enrolled in another investigational drug or investigational medical device study or has participated in an investigational drug or medical device study within 30 days prior to Screening
8. Subject has any condition or situation which, in the investigator's opinion, puts the patient at significant risk, could confound the study results, or may interfere significantly with the subject's participation in the study

   At the Baseline Visit or prior to Randomization, a subject will be excluded from continued participation if the subject has:
9. Subjects that have a mean of the reported 12 hour "average" NPRS responses of < 6 on an eleven-point scale (0 to10) rated over the 5 days prior to the Baseline Visit (as recorded in the electronic Study Diary) in the absence of intolerable side effects as documented in the medical history
10. Subjects with a negative urine test for opioids at Baseline
11. Subjects with a positive Pregnancy test, if applicable
12. Subjects that failed the intrathecal trial during Screening

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Compare the change in Numeric Pain Rating Scale between the IDDS group and the CMM group | Comparisons will be done prior to baseline visit and at 3, 6, 9 and 12 month visits.
  The Numeric Pain Rating Scale (NPRS) is a 0-10 numeric pain rating scale (11 point scale), where a higher scores equates to more pain.
  The primary endpoint for this post-marketing study is the comparison of the NPRS between the IDDS group and the CMM group collected in the Study Diary at various time points.

SECONDARY OUTCOMES:
Compare the change in PROMIS 29 scores between the IDDS group and CMM group | Individual subject scores recorded at baseline visit and at 3, 6, 9 and 12 month visits.
  Compare the subject reported Patient-Reported Outcomes Measurement Information System (PROMIS) 29 between the IDDS group and CMM group. PROMIS 29 assesses pain intensity using a 0-10 numeric rating scale (11 point scale), where a higher score equates to more pain. Other health domains are scored using a Likert scale, where higher scores represent more of the specific domain being measured. The other health domains that are scored are: depression; anxiety; physical function; pain interference; fatigue; sleep disturbance; and ability to participate in social roles and activities.
Comparison of the accrued cost of therapy for pain | Cost of therapy will be obtained at 3, 6, 9 and 12 month visits.
  Compare the accrued cost of therapy for pain control including those related to adverse events, ED visits, cost of medications between the IDDS group and CMM group.
Comparison of other concurrent treatments | Individual subject counts recorded at 3, 6, 9 and 12 month visits will be compared.
  Compare the number of other concurrent treatments performed on each subject between the IDDS group and CMM group.

CONTACTS AND LOCATIONS:
Overall Officials: Jason E Pope, MD, Principal Investigator — Evolve Restorative Center
Locations (1):
- Evolve Restorative Center, Santa Rosa, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deer TR, Pope JE, Hayek SM, Lamer TJ, Veizi IE, Erdek M, Wallace MS, Grider JS, Levy RM, Prager J, Rosen SM, Saulino M, Yaksh TL, De Andres JA, Abejon Gonzalez D, Vesper J, Schu S, Simpson B, Mekhail N. The Polyanalgesic Consensus Conference (PACC): Recommendations for Intrathecal Drug Delivery: Guidance for Improving Safety and Mitigating Risks. Neuromodulation. 2017 Feb;20(2):155-176. doi: 10.1111/ner.12579. Epub 2017 Jan 2. PMID 28042914
- [Background] Deer TR, Hayek SM, Pope JE, Lamer TJ, Hamza M, Grider JS, Rosen SM, Narouze S, Perruchoud C, Thomson S, Russo M, Grigsby E, Doleys DM, Jacobs MS, Saulino M, Christo P, Kim P, Huntoon EM, Krames E, Mekhail N. The Polyanalgesic Consensus Conference (PACC): Recommendations for Trialing of Intrathecal Drug Delivery Infusion Therapy. Neuromodulation. 2017 Feb;20(2):133-154. doi: 10.1111/ner.12543. Epub 2017 Jan 2. PMID 28042906
- [Background] Deer TR, Pope JE, Hayek SM, Bux A, Buchser E, Eldabe S, De Andres JA, Erdek M, Patin D, Grider JS, Doleys DM, Jacobs MS, Yaksh TL, Poree L, Wallace MS, Prager J, Rauck R, DeLeon O, Diwan S, Falowski SM, Gazelka HM, Kim P, Leong M, Levy RM, McDowell G II, McRoberts P, Naidu R, Narouze S, Perruchoud C, Rosen SM, Rosenberg WS, Saulino M, Staats P, Stearns LJ, Willis D, Krames E, Huntoon M, Mekhail N. The Polyanalgesic Consensus Conference (PACC): Recommendations on Intrathecal Drug Infusion Systems Best Practices and Guidelines. Neuromodulation. 2017 Feb;20(2):96-132. doi: 10.1111/ner.12538. Epub 2017 Jan 2. PMID 28042904